CLINICAL TRIAL: NCT03649724
Title: The LUCINDA Trial: LeUprolide Plus Cholinesterase Inhibition to Reduce Neurological Decline in Alzheimer's
Acronym: LUCINDA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Tolmar Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-05020209; R01AG057681-01A1 (NIH)
Record Dates: First submitted 2018-08-22; First posted 2018-08-28 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — luprolide acetate gel depot; Suspensions; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 0.25 ml of sterile normal saline administered subcutaneously / 12 weeks
  Interventions: Drug: Placebo
- Leuprolide (Experimental): Eligard 22.5mg administered subcutaneously / 12 weeks
  Interventions: Drug: Eligard 22.5Mg Suspension for Injection

INTERVENTIONS:
Drug: Placebo — Placebo (0.25 ml normal saline) will be administered subcutaneously once every twelve weeks for 48 weeks.
  Arms: Placebo
Drug: Eligard 22.5Mg Suspension for Injection — Eligard 22.5Mg Suspension for Injection will be administered subcutaneously, in accord with manufacturer's direction, once every twelve weeks for 48 weeks.
  Arms: Leuprolide

SUMMARY:
The LUCINDA Trial is a three-site, phase II, randomized, double-blind, placebo-controlled study of leuprolide acetate (Eligard) in women with Mild Cognitive Impairment or Alzheimer's Disease taking a stable dose of a cholinesterase inhibitor medication like donepezil. Its objective is to assess the efficacy of a 48-week regimen of leuprolide (22.5 mg per 12 weeks) compared to placebo on cognitive function, global function and plasma and neuroimaging biomarkers.

DETAILED DESCRIPTION:
This project aims to re-purpose the safe and well-tolerated gonadotropin-releasing hormone (GnRH) analogue Leuprolide Acetate for use in Alzheimer's Disease (AD). Leuprolide Acetate is currently used in adults for prostate cancer, endometriosis, uterine fibroids and in preparation for in-vitro fertilization, and in children for central precocious puberty. The purpose of this study to confirm and extend results from a prior phase II study (Bowen et al, 2015) which demonstrated that Leuprolide halted cognitive and functional decline in a subgroup of women with mild-moderate AD who were also taking the acetylcholinesterase inhibitor donepezil. Objectives are to replicate, in the same subgroup, Leuprolide's clinical EFFICACY in this prior trial and to add neuroimaging and plasma BIOMARKERS that will help elucidate Leuprolide's likely multiple mechanisms of action in AD. These mechanisms include decreasing levels of Luteinizing Hormone (LH) based on extensive preclinical evidence that decreasing LH preserves cognition and decreases amyloid deposition and tau phosphorylation in animal models of AD, as well as new evidence that GnRH analogues may have anti-inflammatory effects.

ELIGIBILITY:
Inclusion Criteria:

* Female, post-menopausal
* Probable AD or MCI due to AD according to NIA-AA criteria
* Taking a stable dose of a cholinesterase inhibitor such as donepezil/Aricept and dosage likely to remain stable throughout the trial
* MOCA > 11 or blind MOCA > 8 (inclusive) at screening visit
* Hachinski score <5 supporting clinical judgment that dementia is not of vascular origin
* Fluent in English
* has a study partner / caregiver who interacts with the subject for at least 5 hours per week on average and can participate in evaluations

Exclusion Criteria:

* Presence based on exam, history or MRI of significant brain disease other than AD such as schizophrenia, epilepsy, Parkinson's disease or large territory stroke
* Current substance abuse in accord with DSM V criteria
* Significantly depressed (Geriatric Depression Scale > 10)
* Physical or psychological MRI contraindications, or likely unable to tolerate neuroimaging
* Taking other medications known to affect serum sex hormone or gonadotropin concentrations such as estrogen and/or progesterone for hormone replacement therapy, goserelin or danazol
* Presence of significant systemic illness likely to interfere with participation in or completion of the study or to affect study results such as cancer within 5 years (other than non-melanoma skin cancer), autoimmune disease, recent myocardial infarction, signs/symptoms of organ failure based on history, ECG, screening laboratory and/or physical exams
* Receiving other investigational drugs within 30 days or 5 half-lives prior to randomization, whichever is longer

Ages: 60 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog-11) | Baseline, 48 Weeks
  The ADAS-cog-11 consists of 11 tasks measuring the disturbances of memory, language, praxis, attention and other cognitive abilities which are often referred to as the core symptoms of Alzheimer's Disease.

SECONDARY OUTCOMES:
Percent change in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | Baseline, 48 Weeks
  The ADCS-ADL assesses a subject's ability to perform activities of daily living such as eating, walking and bathing.
Alzheimer Disease Cooperative Study Clinical Global Impression of Change (ADCS-CGIC+) | Baseline, 48 Weeks
  The ADCS-CGIC+ uses structured interviews with the subject and his or her caregiver to determine whether there has been a change in the subject's overall level of functioning.
Percent change in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Baseline, 48 Weeks
  The RBANS is a set of tests that measures thinking abilities including memory, language and attention.
Percent change in Burden Inventory | Baseline, 48 Weeks
  The Burden Inventory is a questionnaire that assesses how people sometimes feel when they are taking care of another person.
Percent change in Neuropsychiatric Inventory (NPI) | Baseline, 48 Weeks
  The NPI measures behavioral and emotional symptoms of Alzheimer's Disease.
Change in Brain Magnetic Resonance Imaging (MRI) biomarkers | Baseline, 48 Weeks
  Percent change in volume of AD-related brain regions (hippocampi, ventricles) and hippocampal perfusion measured with Arterial Spin Labeling (ASL) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy A Butler, MD, Principal Investigator — Weill Medical College of Cornell University; James E Galvin, MD, Principal Investigator — University of Miami; Craig S Atwood, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - University of Miami Miller School of Medicine, Boca Raton, Florida
  - Weill Medical College of Cornell University, New York, New York
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The data and resources sharing plan for this project is in accordance with both Weill Cornell and NIH Data Sharing Policies. All raw clinical, genetic, and imaging data from this project will be available upon written request. Deidentified neuroimaging data may be uploaded to one or more of several available data sharing sites designed for this purpose. The final data will be available in acceptable formats such as presentations and publications.
  Research data and results that document and support the study aims will be available after the final results are accepted for publication. The data to be shared will be anonymized and there will be no fees or other restrictions.
Supporting Information: Study Protocol, ICF
Time Frame: Research data and results that document and support the study aims will be available after the final results are accepted for publication.
Access Criteria: Approval from PI

REFERENCES:
- [Background] Butler T, Goldberg JD, Galvin JE, Maloney T, Ravdin L, Glodzik L, de Leon MJ, Hochman T, Bowen RL, Atwood CS. Rationale, study design and implementation of the LUCINDA Trial: Leuprolide plus Cholinesterase Inhibition to reduce Neurologic Decline in Alzheimer's. Contemp Clin Trials. 2021 Aug;107:106488. doi: 10.1016/j.cct.2021.106488. Epub 2021 Jun 22. PMID 34166841
- [Background] Butler T, Glodzik L, Wang XH, Xi K, Li Y, Pan H, Zhou L, Chiang GC, Morim S, Wickramasuriya N, Tanzi E, Maloney T, Harvey P, Mao X, Razlighi QR, Rusinek H, Shungu DC, de Leon M, Atwood CS, Mozley PD. Positron Emission Tomography reveals age-associated hypothalamic microglial activation in women. Sci Rep. 2022 Aug 3;12(1):13351. doi: 10.1038/s41598-022-17315-8. PMID 35922659
- [Background] Wickramasuriya N, Hawkins R, Atwood C, Butler T. The roles of GnRH in the human central nervous system. Horm Behav. 2022 Sep;145:105230. doi: 10.1016/j.yhbeh.2022.105230. Epub 2022 Jul 6. PMID 35809386
- [Background] Butler T, Tey SR, Galvin JE, Perry G, Bowen RL, Atwood CS. Endocrine Dyscrasia in the Etiology and Therapy of Alzheimer's Disease. J Alzheimers Dis. 2024;101(3):705-713. doi: 10.3233/JAD-240334. PMID 39240636
- See also: LUCINDA website — https://jcto.weill.cornell.edu/lucinda

DOCUMENTS (1):
  • Informed Consent Form (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT03649724/ICF_001.pdf